CLINICAL TRIAL: NCT02113462
Title: The Prospective Cohort Study to Investigate the Role of Plasma Triglyceride/High-Density Lipoprotein Cholesterol Ratio To Predict Cardiovascular Outcomes in Chronic Kidney Disease.
Brief Title: Triglyceride/High-density Lipoprotein Cholesterol Ratio in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Associate Professor in Medicine, Gulhane School of Medicine
Other Study IDs: GSM-012014
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Endothelial dysfunction; Inflammation; Insulin resistance; Tg/hdl ratio
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Triglycerides (TG) to High Density Lipoprotein Cholesterol (HDL-C) ratio is a feature of insulin resistance and an independent predictor of cardiovascular risk. The investigators aimed to evaluate the relationship between TG/HDL-C ratio and the endothelial functions in patients with CKD.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) risk is substantially increased in subjects with chronic kidney disease (CKD).The reasons for the elevated risk of CVD in patients with CKD are not fully elucidated. There is not a good prognostic tool for the prediction of increased cardiovascular risk in CKD. A simple, widely available, relatively inexpensive, and generally reproducible marker to predict the CVD risk in subjects with CKD is needed.

The Triglycerides (TG) to High Density Lipoprotein Cholesterol (HDL-C) ratio is a feature of insulin resistance and an independent predictor of cardiovascular risk. No study has been performed so far, to evaluate the role of TG/HDL ratio to predict the CVD risk in patients with CKD.

This study is designed to evaluate the relationship between TG/HDL-C ratio and the endothelial functions in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic kidney disease

Exclusion Criteria:

* taking drugs that may influence endothelial function
* acute infections

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: renal unit
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 months
  The COX analysis was performed in order to establish which covariates were independent predictors of cardiovascular outcomes. Kaplan Meier survival curves are generated to show the impact of the TG/HDL ratio on the cumulative survival of the cohort. The predictive power of the median TG/HDL ratio in each CKD stage for all-cause mortality and cardiovascular events are measured.
Endothelial functions assessed by flow mediated dilatation and serum ADMA measurement | Once in recruitment
  The predictive role of TG/HDL ratio on endothelial functions (ADMA and flow mediated dilatation) is determined by univariate and multivariate analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Sonmez A, Yilmaz MI, Saglam M, Unal HU, Gok M, Cetinkaya H, Karaman M, Haymana C, Eyileten T, Oguz Y, Vural A, Rizzo M, Toth PP. The role of plasma triglyceride/high-density lipoprotein cholesterol ratio to predict cardiovascular outcomes in chronic kidney disease. Lipids Health Dis. 2015 Apr 16;14:29. doi: 10.1186/s12944-015-0031-4. PMID 25885289